CLINICAL TRIAL: NCT02000037
Title: Interest in the Medium Term of an Infrared Reflexotherapy on Overweight or Class I Obese People
Acronym: REFLEX-IR
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The sponsor requested an early termination of the study following insufficient engagement of subjects beyond 12 months of follow-up (initial follow-up was 18 months).
Sponsor: Institut Pasteur de Lille (Other)
Collaborators: Luxomed (Unknown)
Responsible Party: Principal Investigator, Jean-Michel Lecerf, Medical doctor specialized in endocrinology and metabolic diseases, Institut Pasteur de Lille
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2013-A00800-45
Record Dates: First submitted 2013-11-26; First posted 2013-12-03 (Estimated); Last update posted 2022-12-08 (Actual); Status verified 2022-12

CONDITIONS: Assess the Effect of an IR Reflexotherapy on Overweight and Class I Obese People

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Dietary care (Active Comparator): Treatment is composed of a dietary care (with advices on physical activity) given by a professional (dietician of the Nutrition Department of the Institut Pasteur de Lille).
  Interventions: Behavioral: Dietary care
- IR reflexotherapy + dietary care (Experimental): Treatment is composed of :
  * IR reflexotherapy sessions given by a trained professional ;
  * dietary care (with advices on physical activity) given by a professional (dietician of the Nutrition Department of the Institut Pasteur de Lille).
  Interventions: Device: IR Reflexotherapy; Behavioral: Dietary care
- IR Reflexotherapy (Experimental): Treatment is composed of IR reflexotherapy sessions given by a trained professional.
  Interventions: Device: IR Reflexotherapy

INTERVENTIONS:
Device: IR Reflexotherapy — 18 IR reflexotherapy sessions :
  * Once a week for 12 weeks at the beginning of the study
  * Once a week for 3 weeks, 9 months after the beginning of the study
  * Once a week for 3 weeks, 15 months after the beginning of the study
  Arms: IR Reflexotherapy; IR reflexotherapy + dietary care
Behavioral: Dietary care — Dietary consultation 1, 2, 3, 6, 9, 12, 15 and 18 months after the beginning of the study
  Arms: Dietary care; IR reflexotherapy + dietary care

SUMMARY:
The study aim is to Assess the Effect of an IR Reflexotherapy on Overweight and Class I Obese People.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 27 and 35 kg/m2 (included),
* Aged 30 to 60 years old (included),
* Stable weight: no variation of 3 kg in the las 3 months,
* Signed the consent form,
* Able to follow the study,
* Health insured.

Exclusion Criteria:

* History of coronary disease (in the last 6 months),
* Progressive illness at the time of the study (cancer, neurodegenerative disease...),
* Diabetics (treated or not),
* Fasting blood total cholesterol equal or over 2.5 g/L (treated or not),
* Fasting blood triglycerides equal or over 2.0 g/L (treated or not),
* Fasting blood glucose equal or over 1.26 g/L,
* Peripheral neuropathy (polyneuritis, diabetic neuropathy) or central neuropathy (hemiplegia),
* Infectious cutaneous condition or allergies (to the contact point of the device),
* History of stroke,
* Severe heart disease,
* Epilepsy,
* Reduced motility,
* Diagnosed eating disorder,
* Followed a diet in the last 90 days in order to lose weight,
* Took weight loss assistance drug (Orlistat) in the last month or is likely to take one during the study,
* Psychiatric disorder incompatible with the study,
* Mental illness,
* Neurological disorder,
* Chronic somatic disease,
* Addiction or nicotine withdrawal,
* Under psychoactive drug ,
* Alcool consumption over 3 glasses a day,
* Pregnant or breastfeeding women,
* Women that are likely to get pregnant during the study,
* Is unable to understand or follow the protocol
* Is deprived of liberty
* Is under judicial protection

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 87 (Actual)
Dates: Start 2013-10-18 (Actual); Primary Completion 2016-01-28 (Actual); Study Completion 2016-01-28 (Actual)

PRIMARY OUTCOMES:
Weight changes after 12 months compared to a dietary care (associated with physical activity advice) dispensed by a professional. | 12 months

SECONDARY OUTCOMES:
Effect of infrared (IR) reflexotherapy on weight changes. | 3, 12 and 18 months
Effect of IR reflexotherapy combined with a dietary care (and physical activity advises) dispensed by a professional on the weight changes. | 3, 12 and 18 months.
Effect of infrared (IR) reflexotherapy on waist size. | 3, 12 and 18 months
Effect of IR reflexotherapy combined with a dietary care (and physical activity advises) dispensed by a professional on the waist siez. | 3, 12 and 18 months.
Effect of infrared (IR) reflexotherapy on dietary habits. | 3, 12 and 18 months
Effect of IR reflexotherapy combined with a dietary care (and physical activity advises) dispensed by a professional on dietary habits. | 3, 12 and 18 months.
Effect of infrared (IR) reflexotherapy on life's quality (anxiety, depression, physical impact, psychosocial, impact on sexual life, eating well-being, feeling about the dietary care). | 3, 12 and 18 months
Effect of IR reflexotherapy combined with dietary care (and physical activity advises) dispensed by professional on life quality (anxiety, depression, physical impact, psychosocial, impact on sexual life, eating wellbeing, feeling about the dietary care) | 3, 12 and 18 months.
Effect of infrared (IR) reflexotherapy on the salivary cortisol. | 3 months
Effect of IR reflexotherapy combined with a dietary care (and physical activity advises) dispensed by a professional on the salivary cortisol. | 3 months.
Effect of infrared (IR) reflexotherapy on blood pressure and heart rate. | 3 months
Effect of IR reflexotherapy combined with a dietary care (and physical activity advises) dispensed by a professional on blood pressure and heart rate. | 3 months.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Michel LECERF, MD, Principal Investigator — Institut Pasteur de Lille
Locations (1):
- NutrInvest - Institut Pasteur de Lille, Lille, Nord, France